CLINICAL TRIAL: NCT01888861
Title: Evaluating the Effect of Alpha Lipoic Acid on Biochemical Markers, Length of Stay and Other Important Outcomes in Patients Admitted to Intensive Care Units.
Brief Title: Effect of Alpha-lipoic Acid on Biochemical Markers and Important Outcomes in Patients Admitted to Intensive Care Units
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: najmeh hejazi (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, najmeh hejazi, PhD of Nutrition,Shiraz University of Medical Sciences, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 916423
Record Dates: First submitted 2013-06-23; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Oxidative Stress; Inflammation; Malnutrition
Keywords: length of stay in ICU; ventilator free days
MeSH Terms: conditions — Inflammation; Malnutrition | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alpha-lipoic acid (Experimental): the patients in this arm were received 900mg alpha-lipoic acid for 10 days through nasogastric(NG) tube.
  Interventions: Dietary Supplement: alpha-lipoic acid
- placebo (Placebo Comparator): the patients in this arm were received 900mg placebo through NG tube.
  Interventions: Drug: placebo

INTERVENTIONS:
Dietary Supplement: alpha-lipoic acid — the patients in this arm receive 900mg alpha-lipoic acid through NG tube.
  Arms: alpha-lipoic acid
Drug: placebo — the patients in this arm were received 900mg placebo through NG tube.
  Arms: placebo

SUMMARY:
Increasing Reactive oxygen and nitrogen production occurred simultaneously with decreasing serum and intracellular level of antioxidants and enzymes in critical ill patients, which result in increasing ventilator dependency and length of stay in intensive care unit and it also accelerate organ failures in patients. In this double blind clinical trial, the investigators examine effect of alfa-lipoic acid on those patients who admitted to intensive care unit that the investigators expect to stay for more than 7 days in this ward and who have tube feeding and don't have severe liver and kidney failure, AIDS and hepatitis. After randomization of included patients by block randomization the investigators will give 900mg/day alfa-lipoic acid for ten days to treatment group and identical placebo to control group by naso-gastric tube. The purposes of this study are decreasing ventilator dependency period, length of stay in ICU, mortality and decelerate of organ failures.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18;
* expected length of stay more than 7 days;
* using enteral feeding method during admitted to ICU

Exclusion Criteria:

* having the history of autoimmune disease
* severe renal or liver failure
* AIDS,
* hepatitis;
* having severe malnutrition at the admission time;
* having TPN at the admission time in ICU;
* extreme intolerance to enteral feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
length of stay in ICU | day 28
  number of days that patient stay in intensive care unit
mortality | day 28
  percent of mortality
ventilator free days | 10 days
  show by days

SECONDARY OUTCOMES:
sequential organ failure assessment score | 10 days
  determine by SOFA score form
insulin resistance | 10 days
  measure by HOMA calculation equation
malondialdehyde | 10 days
  measure by spectrophotometery
total antioxidant capacity | 10 days
  measure by eliza kit
C reactive protein | 10 days
  measure by nephelometry method
interleukin-6 | 10 days
  measure by eliza kit
Albumin | 10 days
  record from routine lab data of patients in hospital
preAlbumin | 10 days
  by turbidimetric assay
Total lymphocyte count | 10 days
  record from routine lab data of patients in hospital
Mid arm circumference | 10 days
  measure by non flexible meter in mid arm
total protein | 10 days
  record from routine lab data of patients in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Najmeh Hejazi, Ph.D, Principal Investigator — Shiraz University of Medical Sciences,Nutrition department; Zohreh Mazloom, PhD, Study Director — Shiraz University of Medical Sciences, Faculty of Nutrition; Farid Zand, MD, Study Chair — Shiraz University of Medical Sciences, anesthesiology and critical care research center
Locations (1):
- Shiraz University of Medical Sciences, Department of Nutrition, Shiraz, Fars, Iran